CLINICAL TRIAL: NCT06566690
Title: Association Between Sensory Block Level, Oxygen Therapy, and ORi in Varicose Vein Patients Undergoing Spinal Anesthesia: A Correlation Study
Brief Title: The Association Between Sensory Block Level, Oxygen Therapy, and ORi in Varicose Vein Patients Undergoing Spinal Anesthesia (ORi: Oxygen Reserve Index)
Acronym: ORi
Status: Recruiting | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Volkan Alparslan, Asist. Prof. M.D, Kocaeli University
Other Study IDs: 2024-KAEK-02
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hyperoxia; Hypoxia
Keywords: hyperoxia; hypoxia; oxygen therapy; spinal anaesthesia
MeSH Terms: conditions — Hyperoxia; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Addition of ORi monitoring to SpO2 monitoring — Integration of Oxygen Reserve Index (ORi) monitoring into standard SpO2 monitoring

SUMMARY:
The assessment of peripheral capillary oxygen saturation (SpO2) by pulse oximetry has become standard in perioperative care for the detection of hypoxaemia. The oxygen reserve index (ORI) can provide an early warning of deteriorating oxygenation long before a change in SpO2 occurs, reflect the response to oxygen administration, facilitate oxygen titration and prevent unwanted hyperoxia. The combination of ORI with pulse oximetry can help to accurately adjust inhaled oxygen concentration and prevent hypo- and hyperoxaemia. In spinal anaesthesia, neuraxial blockade can cause paralysis of accessory respiratory muscles and theoretically lead to bronchospasm. Therefore, in this study, the investigators planned to perform oxygen saturation monitoring using two modalities. The investigators wanted to investigate the correlation between ORI, SpO2, oxygen therapy and the degree of sensory block.

DETAILED DESCRIPTION:
The assessment of peripheral capillary oxygen saturation (SpO2) by pulse oximetry has become standard in perioperative care for the detection of hypoxaemia. The oxygen reserve index (ORI) can provide an early warning of deteriorating oxygenation long before a change in SpO2 occurs, reflect the response to oxygen administration, facilitate oxygen titration and prevent unwanted hyperoxia. The combination of ORI with pulse oximetry can help to accurately adjust inhaled oxygen concentration and prevent hypo- and hyperoxaemia. In spinal anaesthesia, neuraxial blockade can cause paralysis of accessory respiratory muscles and theoretically lead to bronchospasm. The respiratory effects of neuraxial blockade up to mid-thoracic level are minimal in patients without lung disease. While the intercostal muscles may be paralysed by thoracic block, diaphragmatic function is preserved. Therefore, in this study, the investigators planned to perform oxygen saturation monitoring using two modalities. The investigators wanted to investigate the correlation between ORI, SpO2, oxygen therapy and the degree of sensory block.

ELIGIBILITY:
Inclusion Criteria:

- ASA I-II

Exclusion Criteria:

* Chronic Obstructive Pulmonary Disease (COPD)
* Smoking history of >30 pack-years
* Cancer patients
* Interstitial lung disease patients
* Patients with Body Mass Index (BMI) >30 kg/m²
* Patient refusal of spinal anesthesia
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study aims to include ASA I-II patients aged 18-65 years scheduled for elective varicose vein surgery, with the sample size to be determined by a pilot study
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2026-02-10 (Actual); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of this study is to assess the correlation between the need for oxygen therapy, the ascension of sensory block level, and changes in Oxygen Reserve Index (ORi). | 9 months
  The primary outcome measure of this study is to evaluate the potential correlation between three variables: the need for supplemental oxygen therapy, the cephalad progression of sensory block level, and fluctuations in oxygen reserve index (ORi) values.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Scheeren TWL, Belda FJ, Perel A. The oxygen reserve index (ORI): a new tool to monitor oxygen therapy. J Clin Monit Comput. 2018 Jun;32(3):379-389. doi: 10.1007/s10877-017-0049-4. Epub 2017 Aug 8. PMID 28791567
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28791567/